CLINICAL TRIAL: NCT03709056
Title: A Phase IIb, Randomized, Double-blind, Propofol-controlled, Multi-center Study Evaluating the Efficacy and Safety of HSK3486 for Sedation and Anesthesia in Patients Undergoing Diagnostic Colonoscopy.
Brief Title: A Study Evaluating the Efficacy and Safety of HSK3486
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK3486-203
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Sedation and Anesthesia for Adult Colonoscopy Procedures
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 0.4/0.2mg/kg ，0.5mg/kg/0.15mg/kg (Experimental)
  Interventions: Drug: HSK3486
- Propofol 2.0/1.0mg/kg group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — HSK3486 intravenous (iv) 0.4(0.5) mg/kg for induction, and 0.2 (0.15)mg/kg top-ups for maintenance. 0.3(0.375) mg/kg for induction and 0.15 (0.113)mg/kg for maintenance in adults of 65-70 years old
  Arms: HSK3486 0.4/0.2mg/kg ，0.5mg/kg/0.15mg/kg
Drug: Propofol — Propofol iv 2.0 mg/kg for induction, and 1.0 mg/kg top-ups for maintenance. 1.5 mg/kg for induction and 0.75mg/kg for maintenance in adults of 65-70 years old.
  Arms: Propofol 2.0/1.0mg/kg group

SUMMARY:
A double-blind, randomized, active controlled, multi-center, parallel group study comparing HSK3486 with Propofol, in patients undergoing a colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo a diagnostic or therapeutic colonoscopy;
2. Male or female patients, ASA grade I~III, aged ≥ 18 and≤ 70;
3. Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2;
4. the respiratory rate ≥10 and ≤24, SpO2 when inhaling ≥95%, SBP≥90mmHg, DBP≥60mmHg, HR≥55and ≤100;
5. Patient can understand the procedure of this study and is willing to comply with study requirements. The patient can sign the ICF voluntarily.

Exclusion Criteria:

1. Patients were contraindicated in general anesthesia.
2. Patients with a known sensitivity to propofol, opioids, naloxone, eggs, soy products or a medical condition such that these agents were contraindicated.
3. The patient has some history or evidence of increased risk of sedation or anesthesia, such as cardiovascular disease, respiratory disease, cerebrovascular disease, gastrodintestinal disease and other system disease prior to the screening and/or baseline period.
4. Patients with a history of drug or ethanol abuse with the past 3 months.
5. Patients with respiratory management difficulties.
6. Patients in receipt of any investigational drug within 30 days before screening.
7. Patients in receipt of propofol, opioid , other sedative or anesthetic or analgesics within 72 hours before screening.
8. Abnormal laboratory results consisting of any of the following:

1) neutrophil count≤ 1.5×109/L； 2）platelet≤ 80×109/L； 3）hemoglobin≤ 90 g/L; 4）aspartate aminotransferase≥ 1.5×ULN； 5) serum creatinine≥ 1.2×ULN. 9. Pregnant women or female patients with a positive serum or urine human chorionic gonadotropin pregnancy test at screening or baseline or lactating female patients.

10. Patients with an inability to communicate well with the investigator, or deemed unsuitable according to the investigator (in each case providing a reason)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Success of colonoscopy procedure | from the first dose of the study drug to removal of colonoscope on day 1
  Measured by completion of colonoscopy, no requirement for an alternative sedative or anesthesia drug and no requirement for more than 5 doses of study drug within any 15 minute period.

SECONDARY OUTCOMES:
Time to start of procedure | From first dose of study drug until insertion of colonoscope on day 1
The success rate of the colonoscopy procedure | from the first dose of the study drug to removal of colonoscope on day 1
  The number of patients who successfully completed the colonoscopy procedure accounted for the proportion of all patients in the dose group
Time to fully alert | from the removal of colonoscopy procedure, until the first of three consecutive MOAA/S scores of 5 on day 1
Time to discharge | from the removal of colonoscopy procedure, until the first of three consecutive Aldrete scores of more than or equal to 9 on day 1
Application of study drug and alternative medication | during the colonoscopy procedure on day 1
  total dosages of study drug and alternative medication

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - West China Hospital, Sichuan University, Changde
  - The Second Xiangya Hospital of Central South University, Changsha
  - The Third Xiangya Hospital of Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - Shanghai Fengxian District Central Hospital, Shanghai
  - The second Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - General Hospital of Ningxia Medical University, Yinchuan